CLINICAL TRIAL: NCT00816218
Title: Molecular Mechanisms of Endothelial Dysfunction in Type 2 Diabetes Mellitus
Brief Title: Molecular Mechanisms of Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 012-5014-401
Record Dates: First submitted 2008-12-15; First posted 2009-01-01 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pioglitazone (Experimental): Fifty type 2 diabetic patients (25 diet-treated and 25 treated with diet plus sulfonylurea) will have pioglitazone, 45 mg daily; added to their therapeutic regimen. All patients will be closely monitored and, in addition to periodic contacts and clinical visits, metabolic and vascular parameters will be assessed at the beginning and after 3 and 6 months of therapy. Euglycemic hyperinsulinemic clamp with muscle biopsies will be performed at the beginning and after 6 months of treatment.
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — pioglitazone, 45 mg daily
  Other Names: Actos

SUMMARY:
This project is designed to evaluate the molecular mechanisms involved in the early development of endothelial dysfunction in type 2 diabetic patients. The investigators intend to correlate increases in insulin signaling pathway activity following pioglitazone therapy with improvements in nitric oxide synthase expression in skeletal muscle. In addition, the investigators will evaluate vascular responses and in vivo nitric oxide release during administration of acetylcholine and nitroprusside in patients with type 2 diabetes. Enhanced knowledge of the molecular mechanisms responsible for endothelial dysfunction, an early abnormality in the pathogenesis of atherosclerosis, is critical before novel therapies to arrest or delay the appearance of cardiovascular complications in diabetes can be developed.

The investigators intend to recruit fifty type 2 diabetic patients treated with diet alone or diet plus sulfonylureas or meglitinides and add Pioglitazone (45 mg), an insulin sensitizer, for 6 months. In addition to assessment of clinical and metabolic parameters, insulin sensitivity and brachial artery and skin microcirculatory responses to acetylcholine and nitroprusside in combination with simultaneous determination of nitric oxide release will be documented before, 3 and 6 months after Pioglitazone therapy is initiated. Circulating levels of markers of endothelial damage (VCAM, ICAM, selectins), inflammation (C-reactive protein and interleukins), increased coagulability (PAI-1) as well as lipids and apolipoproteins will measured during the study. Skeletal muscle biopsies will be performed during the euglycemic insulin clamp before and 6 months after therapy for measurements of NO synthase activity and key elements of the insulin signal transduction pathway involved in the regulation of glucose metabolism (IRS-1, PI-3 kinase, PI-3 kinase associated with IRS-1 and the mitogenesis MAP-kinase.

Type 2 diabetes confers a substantial increase in the risk of cardiovascular disease. This is believed to be due, in part, to endothelial dysfunction, which correlates closely with impaired vascular responsiveness. Our study will clarify further the extent to which resistance to insulin action and impaired nitric oxide release from endothelial cells are interrelated. We also expect to demonstrate that insulin sensitizers (pioglitazone) can help to restore normal endothelial function, and ultimately prevent/delay the appearance of vascular disease in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Specific Aims

To test the global hypothesis that increases in insulin signaling through either PI-3-kinase or MAP kinase pathways correlate with improvements in NO production or NOS expression in skeletal muscle following pioglitazone therapy, we will determine whether 6 months of Pioglitazone therapy:

i. Increases the activities of muscle NO synthase, IRS-1, PI-3 kinase, PI3-kinase associated with IRS-1 and/or MAP-kinase ii. Improves brachial arterial endothelial function In addition, we will determine whether 6 months of pioglitazone therapy improves abnormal cardiovascular disease risk factors in type 2 diabetic patients by documenting the effects of the drug on plasma lipoprotein profile and on circulating levels of markers of hypercoagulability, inflammatory and endothelial damage.

Experimental Plan Subjects. Adult type 2 diabetic individuals ranging from 18-65 yrs, with BMI between 24 and 37 kg/m2 and mean hemoglobin A1c levels equal to 6.5 and 9.0% will be studied. A total of 50 subjects will be recruited. There are over 8,000 type 2 diabetic patients under treatment at the TDI with a total of approximately 90,000 visits per year registered in the year 2000. As the main source of diabetes care and education to a population of predominantly Hispanic Americans, the TDI also is responsible for periodic screening in the community. Thus, we do not anticipate any problems in recruiting 50 subjects required for the present study. All patients will be normotensive, free of significant medical problems other than diabetes, and either on diet alone or diet plus sulfonylurea (or meglitinides) therapy. Subjects who have received or are receiving treatment with a thiazolidinedione (TZD) will be excluded. We previously have shown that sulfonyureas have no direct insulin sensitizing effect.

Research Design. General Approach. An open-label prospective clinical trial including 50 type 2 diabetic patients (25 diet-treated and 25 treated with diet plus sulfonylurea) will have pioglitazone, 45 mg daily; added to their therapeutic regimen. All patients will be closely monitored and, in addition to periodic contacts and clinical visits, metabolic and vascular parameters will be assessed at the beginning and after 3 and 6 months of therapy. Euglycemic hyperinsulinemic clamp with muscle biopsies will be performed at the beginning and after 6 months of treatment.

Subject Recruitment. Potential volunteers will be invited for a screening visit (Visit 1) during which subjects will be instructed in English (with Spanish translation when appropriate) about the nature of the study, eligibility criteria and required commitments, as well as the potential risks and benefits anticipated for each individual and for the community in general. Written informed consent for participation in the clinical trial from individuals thought to be eligible to participate will be obtained at Visit 1.

At Visit 1 a complete medical history (including a list of current medications, reproductive status and menstrual history for females), physical examination (including height and weight), and vital signs will be obtained. Three consecutive blood pressure measurements will be performed in the sitting position using an automated arm cuff and only individuals with a blood pressure less than 140/90 mmHg will be considered eligible. A urinalysis will be performed and blood will be drawn after an overnight fast for measurement of complete blood count (hematocrit, white cells and platelets), plasma glucose, free T4 and TSH; SMA 20, lipid profile; hemoglobin A1c levels (HbA1C); free fatty acids, insulin and C-peptide concentrations and for a pregnancy test (females only). An EKG also will be performed. All diabetic patients who are deemed healthy and meet eligibility criteria (see below) based upon physical exam, medical history and screening laboratory tests will be invited to participate in the study.

Subjects must meet all of the following criteria: 1) male or female 18-65 years of age; 2) type 2 diabetes based on the American Diabetes Association criteria; 3) HbA1c = 6.5-9.0% while on diet alone or diet plus sulfonylurea (or meglitinides) therapy; 4) no history of thiazolidinediones, insulin, ACE inhibitor or AII-receptor blockade therapy; 5) taking no medications known to affect glycemic control or endothelial function, unless the medication has been stable for at least 3 months; 6) blood pressure equal or below 140/90 mmHg; 7) not pregnant and willing to take appropriate contraceptive measures if capable of becoming pregnant; 8) serum creatinine below 1.7 mg/dl in female and 1.8 mg/dl in males; 9) ALT or AST less than 2 times the upper limit of normal for the laboratory and absence of clinical signs or symptoms of liver disease; 10) hematocrit > 34% in females and >35% in males; 11) normal thyroid function; 12) no evidence of coronary heart disease (by history or EKG) or moderate to severe congestive heart failure (NY Heart Association Cardiac Class III or IV); 13) no history or the presence of any clinically significant or unstable medical condition that makes the subject unlikely to complete the study in the opinion of the PI; and 14) absence of any condition or situations which would preclude adherence and completion of the protocol; 15) the ability to give voluntary informed consent. All clinical laboratory analyses for this trial will be performed at the central laboratory at the University of Texas Health Science Center in San Antonio. All research analytical determinations will be performed in the laboratories of the Diabetes Division. Eligible subjects will return one week after Visit 1 for a second visit (Visit 2), a subject number will be assigned, and a nutritional assessment by a dietitian will be performed. A morning urine specimen will be collected for the determination of microalbumin-to-creatinine ratio. Patients also will have baseline determinations of circulating plasminogen activator inhibitor PAI-1, endothelin-1, VCAM, ECAM, p-selectin and e-selectin (markers of endothelial damage), C-reactive protein and interleukins (markers of inflammation); PAI-1 (marker o hypercoagulable state); plasma lipids (total HDL/LDL cholesterol and triglycerides), as well as LDL and HDL particle size, and apolipoproteins A1, B and C-III. All personal data, anthropometric measurements (height, weight, waist-to-hip ratio), dietary history, vital signs and clinical findings will be recorded in a confidential master file.

Euglycemic Insulin Clamp with Muscle Biopsies. The degree of insulin resistance will be estimated with the euglycemic hyperinsulinemic clamp technique (23) using an insulin infusion rate (80 mU/m2.min), as previously described (24). Briefly, one week after completion of the screening visit 2 (Visit 3), patients will report to the Clinical Research Unit at 8:00 AM after a 10-12 hour overnight fast. Catheters will be inserted into a peripheral vein (for infusion of all test substances) and into a retrograde hand vein (for blood sampling), which will be placed in a heated box (750 C). At time t = -120 minutes, a percutaneous biopsy of the vastus lateralis muscle will be performed under local anesthesia as previously described (25). The subject then will be allowed to rest in bed for 60 minutes. At time t = -30 min to 0 min baseline blood samples will be obtained. At time = 0 min, insulin will be infused at 80 mU/m2.min for 180 minutes to raise the plasma insulin concentration to approximately 120 µU/ml to examine peripheral tissue (muscle) sensitivity to insulin. During the insulin clamp, a small amount of blood (0.5 ml) is withdrawn every 5 minutes from the arterialized venous blood (heated box technique) to determine plasma glucose concentration. When the plasma glucose concentration declines to 100 mg/dl a variable infusion of 20% dextrose is appropriately adjusted to maintain the plasma glucose concentration constant at this level (±5%). The rate of exogenous glucose infusion will be averaged during the last 60 minutes to provide a quantitative measure of insulin-mediated (primarily muscle) total glucose disposal. Insulin infusion will be stopped and the study will be terminated at t = 180 minutes. Patients will be observed for an additional 90 minutes after consuming a meal and they will be allowed to leave after plasma glucose is stable.

Vascular Studies. Subjects will be asked to return to the Clinical Research Unit one week after the euglycemic insulin clamp for vascular studies (Visit 4). Change in forearm blood flow following brachial artery infusion of acetylcholine (endothelial NO-dependent) and sodium nitroprusside (endothelial-independent) will be used to assess the arterial vasodilatory response to physiological stimuli. All test substances will be infused into the non-dominant arm. After local skin anesthesia with lidocaine, a 20-gauge needle attached to an arterial line (Arrow International, Erding, Germany) will be used to cannulate the brachial artery. A pressurized 0.9% saline solution bag will be connected to the arterial line, and a constant drip will be started at t = -60 min to keep the arterial line patent throughout the study. Subjects will then be allowed to rest for 60 minutes. At time t = -5 min, five consecutive measurements of forearm blood flow will be performed using a mercury strain gauge plethysmography (Hokanson Plethysmograph, Model EC4, Hokanson, Bellevue, WA), combined with a rapid cuff inflator. Test substances will be infused according to a variation of the original design of Bergholm et al, as follows. After completion of baseline measurements, an intra-brachial infusion of sodium nitroprusside at 3 microg/min will be started and continued for 12 minutes (the last 6 minutes are used to establish the local vascular effect of sodium nitroprusside). At time t = 12 min, the infusion rate of sodium nitroprusside is increased to 10 microg/min and the infusion continued for an additional 6 minutes. At time t = 18 min, the sodium nitroprusside infusion is stopped and 2 ml of blood is withdrawn to clear the arterial line. Saline is then infused for 30 minutes and at time t = 48 min, an intra-brachial infusion of acetylcholine at a constant rate of 15 microg/min is started and continued for 8 minutes (the last 6 minutes are used to establish the local vascular effect of acetylcholine). At time t = 54 min, the infusion rate of acetylcholine is doubled to 30 microg/min and the infusion continued for and additional 6 minutes. Forearm blood flow is measured five consecutive times during the last 3 minutes of each intra-brachial infusion period, i.e., at time t = 9-12 min and t = 15-18 min, respectively during the low and high nitroprusside dose, and at time t = 51-54 min and t = 57-60 min, respectively during the low and high acetylcholine dose. At time t= 60 min, the acetylcholine infusion is stopped and the study terminated. At the end of the experiment the arterial line is removed and compression to the area applied for 10 minutes. The radial pulse is verified every 5 minutes during the 30-min period after the experiment is terminated, before subjects are allowed to leave. Subjects will be contacted within 24 hrs and 1week after completion of the study to ascertain that there have been no complications.

Upon completion of baseline metabolic and vascular studies patients will be started on pioglitazone, 30 mg per day (Visit 6). Patients will be asked to continue with their previous medical regimen and will be followed by the PI/nursing team at the Texas Diabetes Institute. All participants will be contacted weekly by phone to ascertain that there are no adverse events during the initiation period of 4 weeks, at which time the dose of pioglitazone will be increased to 45 mg per day. All patients will be required to return for office visits at 6 weeks intervals during the entire 6 months of the study (Visits 7-10). All available records of capillary blood glucose, adverse events and other major events will be collected and added to a confidential file under the patients' assigned number. Office visits every six weeks are intended to review patients' interim medical history to document adverse events, to emphasize adherence to the medical regimen, to obtain blood for laboratory determinations, and record vital signs, body weight, neurologic and fundoscopic findings. Blood and urine measurements similar to those in Visit 2 also will be obtained. Metabolic and vascular studies similar to those described above (Visits 3,4,5) before the initiation of pioglitazone therapy will be performed again at 3 and 6 months (Visits 8 and 10) and insulin clamps with muscle biopsies will be repeated at the end of the 6 month period (Visit 10). Patients will be discontinued from the study program for any of the following reasons: 1) the principal investigator decides that the subject should be withdrawn, either because of serious adverse events or clinically significant laboratory abnormalities; 2) the subject requests that he/she be withdrawn; 3) the subject becomes pregnant during the study; and 4) the subject is non-compliant with study guidelines, recommendations, and for the treatment regimen. Early termination at any time will be accompanied by collection of data as outlined in Visit 10. Any patient who is withdrawn from the study will be followed for as long as necessary to establish a stable therapeutic program.

Laboratory Tests. Measurements of fasting plasma glucose (Beckman Glucose Analyzer), HbA1c (32) insulin (33) and C-peptide (34) by radioimmunoassay, and free fatty acids by HPLC (35) will be performed in the principal investigator's laboratory at the Texas Diabetes Institute, as previously described. Assays for VCAM and ICAM (3), p-Selectin and s-Selectin (4), PAI-1 and endothelin-1 (36), and plasma lipids by MRS (37) and apolipoproteins (38) will be performed in the laboratories of the Diabetes Division at the University of Texas Health Science Center. Measurements of IRS-1 thyrosine phosphorylation, PI-3 kinase activity and association of PI-3 kinase with IRS-1 also will be performed in the Diabetes Division laboratory.

Sample Size and Data Analysis Methods. We will perform correlation analyses to examine the relationships between the increment in skin and forearm blood flow following acetylcholine infusion and the improvements in plasma hemoglobin A1c levels and whole body insulin sensitivity before and after pioglitazone therapy using ANOVA with repeated measures over time. We anticipate that pioglitazone treatment will improve glycemic control and tissue insulin sensitivity and that the improvements in hemoglobin A1c and insulin action will be closely related to improvements in acetylcholine-stimulated increments in skin and forearm blood flow. Changes in insulin sensitivity (insulin clamp data), insulin signaling pathways activity, nitric oxide production in vivo, endothelial function, FPG and HbA1c will be compared. Further, we anticipate that plasma levels of endothelial damage markers (ICAM/VCAM), p-Selectin, s-Selectin and PAI-1 and inflammatory markers (C-reactive protein and interleukins), which are elevated in diabetic patients, will be reduced following pioglitazone, and that the reduction will correlate with the improvements in skin and muscle endothelial function. We also expect to observe an improvement in the plasma lipid profile, especially triglycerides and free fatty acids after pioglitazone treatment. Similar correlations between improved endothelial-independent blood flow (nitroprusside-stimulated) following pioglitazone treatment and enhanced insulin sensitivity, glycemic control, nitric oxide production and insulin signaling pathways will also be performed. We expect that improved insulin sensitivity (insulin clamp) and increased NO production in vivo following pioglitazone treatment will be closely related to enhanced IRS-1 tyrosine phosphorylation and total IRS-1 associated PI-3 kinase activity, which we previously have shown to be markedly impaired in type 2 diabetic individuals (39). In contrast, we expect that the MAP-kinase (mitogenic) pathway, which regulates vascular smooth muscle cell growth/proliferation and which we have shown to be normal or upregulated in type 2 diabetics, may be inhibited following pioglitazone treatment. It would be of great pathogenic significance if reduction in the MAP kinase activity correlated with the improved endothelial function following pioglitazone therapy.

The sample size calculation was based upon the changes in forearm blood flow in response to acetylcholine and sodium nitroprusside in normal and diabetic subjects during preliminary studies and from previously published studies by Caballero et al (10). The pooled standard deviation for changes from baseline to endpoint in forearm blood flow (ml/100gr per min) in our laboratory is 1.20. In order to detect with 90% power a difference in forearm blood flow in response to these physiologic agents before and after 6 months of pioglitazone therapy, 40 completed patients are required. Assuming a dropout rate of approximately 20%, 50 diabetic patients must be recruited to obtain 40 completers. Based on the laser Doppler skin blood flow measurements, we have an 80% chance of showing an improvement of ~50% in skin blood in response to physiologic stimuli (from 65% to 100%) following pioglitazone therapy. Thus, we will have more than sufficient diabetic individuals to detect statistically significant changes in skin and muscle blood flow.

ELIGIBILITY:
Inclusion Criteria:

1. male or female 18-65 years of age;
2. type 2 diabetes based on the American Diabetes Association criteria;
3. HbA1c = 6.5-9.0% while on diet alone or diet plus sulfonylurea (or meglitinides) therapy;
4. no history of thiazolidinediones, insulin, ACE inhibitor or AII-receptor blockade therapy;
5. taking no medications known to affect glycemic control or endothelial function, unless the medication has been stable for at least 3 months;
6. blood pressure equal or below 140/90 mmHg;
7. not pregnant and willing to take appropriate contraceptive measures if capable of becoming pregnant;
8. serum creatinine below 1.7 mg/dl in female and 1.8 mg/dl in males;
9. ALT (SGTP) or AST (SGOT) less than 2 times the upper limit of normal for the laboratory and absence of clinical signs or symptoms of liver disease;
10. hematocrit > 34% in females and >35% in males;
11. normal thyroid function;
12. no evidence of coronary heart disease (by history or EKG) or moderate to severe congestive heart failure (NY Heart Association Cardiac Class III or IV);
13. no history or the presence of any clinically significant or unstable medical condition that makes the subject unlikely to complete the study in the opinion of the PI; and
14. absence of any condition or situations which would preclude adherence and completion of the protocol;
15. the ability to give voluntary informed consent.

Exclusion Criteria:

1. Subjects were excluded from study if they had ever received insulin, metformin, TZDs, exenatide or DPP IV inhibitor.
2. All subjects were free of cardiovascular, renal or major organ disease, as determined by medical history, physical examination, screening blood chemistries, complete blood cell count, and electrocardiogram.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2003-03; Primary Completion 2006-07 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Vascular Endothelial Function | at 3 , 6 and 9 months post-therapy
  Brachial arterial dilation and blood flow

SECONDARY OUTCOMES:
Insulin Resistance | Basal and 9 months
  Inmsulin-mediated glucose disposal

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Cersosimo, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Derived] Coletta DK, Sriwijitkamol A, Wajcberg E, Tantiwong P, Li M, Prentki M, Madiraju M, Jenkinson CP, Cersosimo E, Musi N, Defronzo RA. Pioglitazone stimulates AMP-activated protein kinase signalling and increases the expression of genes involved in adiponectin signalling, mitochondrial function and fat oxidation in human skeletal muscle in vivo: a randomised trial. Diabetologia. 2009 Apr;52(4):723-32. doi: 10.1007/s00125-008-1256-9. Epub 2009 Jan 24. PMID 19169664